CLINICAL TRIAL: NCT07159321
Title: Frailty and Health-related Quality of Life in Older Women With Breast Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shorouq Alaaeldin Abdelaziz Elsayed, assistant lecturer of Geriatric medicine, Ain Shams University
Other Study IDs: palliative 2025-6
Record Dates: First submitted 2025-07-14; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Females; Frailty
MeSH Terms: conditions — Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Females aged 60 years and older, who are newly diagnosed with pathologically proven breast inva
  Interventions: Other: Comprehensive geriatric assessment; Other: European Organization for Research and Treatment-Quality of life questionnaire; Other: Clinical Frailty Scale

INTERVENTIONS:
Other: Comprehensive geriatric assessment — Functional status will be evaluated using Activities of Daily Living (ADL) (assessing bathing, dressing, toileting, transferring, eating, and continence; Katz, 1970) and Instrumental ADL (IADL) (assessing shopping, cooking, medication management, phone use, housework, laundry, transportation, and finances; Lawton & Brody, 1969). Nutritional status will be measured via the Mini-Nutritional Assessment-Short Form (MNA-SF) (Arabic version; Abd-Al-Atty et al., 2012), a 6-item tool (appetite, weight loss, mobility, illness, neuropsychological issues, BMI) scored 0-14, classifying patients as well-nourished (≥12), at risk (8-11), or malnourished (0-7; Rubenstein et al., 2001). Cognition will be assessed using the Saint Louis University Mental Status (SLUMS) exam (Arabic version; Abdelrahamn et al., 2014), a 30-point test evaluating calculation, orientation, memory, fluency, and visuospatial function, with dementia thresholds at <20 (<12 years education) or <21 (≥12 years; Tariq et al., 2006).
Other: European Organization for Research and Treatment-Quality of life questionnaire — Quality of life assessment by European Organization for Research and Treatment-Quality of life questionnaire and breast cancer-specific module (EORTC QLQ-C30)and QLQ-BR23)
  EORTC QLQ-C30 is a validated tool designed to measure cancer patients' physical, psychological and social functions. It consists of 30 items measuring Global Health status (2 items), Functional scales (15 items) and Symptoms scales/items (13 items). Items were measured using a 4-point Likert Scale ranging from Not at all (1) to Very much (4).
  EORTC-BR23 consists of 23 items which measure two main scales "Functional Scale (8 items) and "Symptoms scales (15 items). Items measured using 4-point Likert Scale ranging from Not at all (1) to Very much (4).
Other: Clinical Frailty Scale — Frailty will be assessed using the Clinical Frailty Scale (CFS), a validated and widely used tool developed by (Rockwood et al., 2005). The CFS is a 9-point ordinal scale that categorizes older adults based on their level of physical fitness, functional independence, and comorbidities, ranging from 1 indicate very fit to 9 indicate terminally ill. Participants were evaluated by trained clinicians based on their clinical judgment, incorporating information from patient interviews. The scale provides a practical and reliable measure of frailty in geriatric populations and has demonstrated strong predictive validity for adverse health outcomes including hospitalization, institutionalization, and mortality.

SUMMARY:
This study addresses a critical gap in the care of older women with breast cancer, a population often underrepresented in clinical research despite their increased vulnerability to treatment-related complications. By examining the relationship between frailty and health-related quality of life (QOL), the study aims to provide evidence-based insights into how geriatric assessments can guide personalized treatment decisions, ensuring that therapeutic benefits outweigh risks. Given that older adults prioritize QOL over survival gains, understanding the impact of frailty on their well-being can help clinicians optimize care plans, reduce adverse outcomes, and improve overall patient-centered outcomes. The findings may also inform the integration of routine geriatric assessments in oncology practice, ultimately enhancing the management of older cancer patients in resource-limited settings like Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 60 years and older
* Newly diagnosed with pathologically proven breast invasive ductal or lobular carcinoma

Exclusion Criteria:

* History of cognitive impairment or psychiatric disorders
* Delirium during assessment using the Confusion Assessment Method (CAM test)
* Initiation of chemotherapy before the baseline assessment
* Severe hearing or visual impairment preventing completion of assessment
* Other malignancies (second primary)
* Other breast malignancies (e.g., sarcoma)
* End-organ failure (e.g., renal failure, liver cell failure)

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: older females; 60 years old or older, diagnosed with breast cancer before receiving chemotherapy will be recruited from the clinical oncology department, Ain Shams university hospitals.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Quality of life measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 and 23. | 6 months
  Health-related quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) together with the Breast Cancer-Specific Module. Both instruments generate scores ranging from 0 to 100. For functional domains and global health status, higher scores indicate better quality of life, whereas for symptom domains, higher scores indicate more severe symptoms and worse outcomes at baseline and 6 months.

SECONDARY OUTCOMES:
change in Frailty status as assessed by clinical frailty scale | 6 months
  Frailty assessed via Clinical Frailty Scale (CFS) at baseline and 6 months. The Clinical Frailty Scale (CFS) is a 9-point scale ranging from 1 (very fit) to 9 (terminally ill). Higher scores reflect increasing levels of frailty and are associated with poorer outcomes, while lower scores indicate better physical reserve and functional status.

IPD SHARING:
Plan to Share IPD: Undecided